CLINICAL TRIAL: NCT04764734
Title: A Validation Study of the NightOwl Home Sleep Apnea Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ectosense NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NightOwl-02
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Single Group will undergo both gold standard polysomnography (PSG) and NightOwl Sleep Apnea Test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PSG and NightOwl (Experimental): During the study, for each execution day, all patients that have been scheduled for a PSG will be presented with the informed consent form. All recruited patients shall be a part of the study during which they wear the NightOwl Sensor while undergoing the PSG exam.
  Interventions: Device: NightOwl

INTERVENTIONS:
Device: NightOwl — The NightOwl is a finger-mounted home sleep apnea testing device

SUMMARY:
The objective of this study is to evaluate the performance of a miniaturized sleep apnea test, called NightOwl. The system consists of a sensor placed on the fingertip and a cloud-based analytics software. The sensor acquires accelerometer and photoplethysmographic data. The software derives actigraphy from the former, and blood oxygen saturation and peripheral arterial tone (PAT), among other features, from the latter. In order to assess NightOwl's performance, the investigators will compare the apnea hypopnea index (AHI) estimate, defined as the number of respiratory events per hour of sleep, derived by the NightOwl system, to the apnea-hypopnea index (AHI) obtained from manual analysis of the polysomnography (PSG), which is the gold standard for sleep apnea diagnosis. This study will be performed in a sleep lab environment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with an indication for an in-lab polysomnography

Exclusion Criteria:

* Intellectually disabled people

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-20 (Actual); Primary Completion 2022-09-05 (Estimated); Study Completion 2022-09-10 (Estimated)

PRIMARY OUTCOMES:
The Evaluation of the Level of Agreement (Classification Accuracy) Between Patient Categorization | Through study completion, an average of 1 month.
  The evaluation of the level agreement (classification accuracy) between patient categorization (into sleep apnea severity categories) obtained by the NightOwl and those obtained by the PSG. This measure is calculated by dividing the number of participants on which both NightOwl and the PSG agree on the sleep apnea severity category by the total number of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jagdeep Bijwadia, MD MBA, Principal Investigator — SleepMed RX
Locations (4):
- United States (4):
  - Coral Springs Laboratory, Coral Springs, Florida
  - United Sleep Diagnostics Hollywood Laboratory, Hollywood, Florida
  - Miami Lakes Laboratory, Miami Lakes, Florida
  - United Sleep Diagnostics Pembroke Pines Laboratory, Pembroke Pines, Florida

IPD SHARING:
Plan to Share IPD: No